CLINICAL TRIAL: NCT00971581
Title: Safety, Tolerability and Efficacy of FDC Ketoprofen + Omeprazole in Patients With Rheumatological Conditions With History or Who Are at Risk of Developing NSAID Associated Benign Gastric Ulcers, Duodenal Ulcers and Gastroduodenal Erosions
Brief Title: Safety, Tolerability and Efficacy Study With a Fixed-Dose Combination (FDC) Ketoprofen Plus Omeprazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KETOM_L_04584
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

ARMS (1):
- FDC KETOPROFEN+OMEPRAZOLE (Experimental): One capsule of Ketoprofen 200 mg + Omeprazole 20 mg FDC once daily Treatment duration: 4 weeks
  Interventions: Drug: FDC KETOPROFEN+OMEPRAZOLE

INTERVENTIONS:
Drug: FDC KETOPROFEN+OMEPRAZOLE — Ketoprofen + Omeprazole FDC once daily for 4 weeks

SUMMARY:
Primary Objective:

To confirm the safety and tolerability of the fixed dose combination of a Non-Steroidal Anti-Inflammatory Drug (NSAID), ketoprofen, associated to a Proton Pump Inhibitor (PPI), omeprazole, in Mexican patients.

Secondary Objective:

To confirm the efficacy of the combination:

* Relief of pain (Visual Analyzed Score (VAS))
* Patients global assessment of disease activity, scored as a scale of 1 (no limitation of normal activities) to 5 (inability to carried out all normal activities)

ELIGIBILITY:
Inclusion criteria:

* Adults suffering from chronic inflammatory conditions, in particular, rheumatoid polyarthritis, ankylosing spondylitis (or related syndromes, such as, Reiters syndrome, psoriatic arthritis,) with a previous history or who are at risk of developing NSAID associated benign gastric ulcers, duodenal ulcers and gastroduodenal erosions in whom continued treatment with NSAIDs is necessary.
* Presenting at the inclusion visit an acute episode of recent onset (<48 hours) defined by average pain within the last 24 hours >=50 mm on the Visual Analogue Scale (VAS).

Exclusion criteria:

* Hypersensitivity to ketoprofen or to omeprazole or to another proton-pump inhibitor or to any of the excipients.
* Last trimester of pregnancy.
* History of asthma induced by administration of ketoprofen or similar acting substances, such as other non-steroidal anti-inflammatory agents (NSAIDs) or acetylsalicylic acid.
* Gastrointestinal disorder or surgery leading to impaired drug absorption.
* Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion would endanger a subject if they were to participate in the study.
* Serious blood coagulation disorder including use of systemic anticoagulants.
* Positive test result for H. pylori at screening.
* Recent endoscopy showing any gastric or duodenal ulcer at least 3 mm in diameter with depth.
* Severe hepatic failure.
* Severe renal failure.
* Severe heart failure.
* Patients with asthma associated with chronic rhinitis, chronic sinusitis and/or nasal polyposis.
* Active peptic ulcer.
* Gastrointestinal bleeding, cerebrovascular bleeding or other active bleeding.
* Alcohol consumption or drug abuse.
* Concomitant use with St. Johns wort or atazanavir sulphate.
* Concomitant use of the following medications:

  * NSAIDs including cyclooxygenase-2 selective inhibitors
  * Salicylates
  * Corticosteroids
  * DMARDs
  * Antacids
  * Histamine H2 receptors
  * Misoprostol
  * Other PPI
  * Sucralfate
  * Anticoagulants: Anti-platelet agents and selective serotonin reuptake inhibitors (SSRIs)
  * Lithium:
  * Methotrexate (at doses above 15 mg/week):
* Screening laboratory value for ALT, AST >2 times the upper limit of normal.
* Other than noted specifically, any screening laboratory value that is clinically significant in the investigator's opinion and would endanger a subject if they were to participate in the study.
* History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.
* Participation in any study of an investigational treatment in the 8 weeks before screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To confirm the efficacy of the combination | From the start to the end of the study (D 0 to D 28)
Incidence of dyspeptic symptoms: epigastric pain, dyspepsia, nausea | At Day 10

SECONDARY OUTCOMES:
Incidence of dyspeptic symptoms: epigastric pain, dyspepsia, nausea | At Day 0, Day 4 & Day 28
Incidence of complications (perforations, ulcers, bleeding) and Incidence of fecal occult blood positivity | At study termination (Day 28)
Improvement of pain (VAS) | At study termination (Day 28)
Incidence of moderate to severe abdominal symptoms and GastroIntestinal Adverse Event leading to withdrawal | From the start to the end of the study (D 0 to D 28)
Patient's global assessment of disease activity, scored as a scale of 1 (no limitation of normal activities) to 5 (inability to carried out all normal activities) | At study termination (Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico